CLINICAL TRIAL: NCT03496558
Title: Model of Variability of the Lipid Profile in Pregnant Women and Its Relationship to lactogénesis
Acronym: PLELACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, María José Aguilar Cordero, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 28/06/2017 UGR
Record Dates: First submitted 2017-07-06; First posted 2018-04-12 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Pregnant Woman With Single Pregnancy; Pregnant Woman With no Assisted Reproduction
Keywords: lactogenesis, pregnant, TG, lipidic profile, breastfeeding.
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 pregnant women with a history of risk (Experimental)
  Interventions: Other: Variability of the lipid profile in pregnant women
- 150 healthy pregnant women (No Intervention)

INTERVENTIONS:
Other: Variability of the lipid profile in pregnant women — The women participants will be divided into two groups. Group 1 comprised of healthy women and group 2 by pregnant women with a history of risk. A personal, family history and a detailed medical history will be taken in each group. We will proceed to see all possible variables that influence the level of biomarkers (lipids and prolactin).
  At least 60 healthy pregnant women and 60 pregnant women with a history of risk (20 for each risk) x 2 series (three years) will be tried, a total of 240-300 women to whom 5 analytical tests would have to be performed.
  Arms: 150 pregnant women with a history of risk

SUMMARY:
The project that is presented to the ethical committee, from the initial program called BECOME (Behavior of biomarkers (lipid profile and prolactin) during pregnancy and lactation through a biological multi-paradigm model), which already requested and obtained the Suitability dated April 28, 2015. Based on it, the development of the current project will be the historical memory of FPU Research Fellow (October 2016) The determination of the lipid profile in pregnancy is performed through blood tests in each of the quarters.

A prospective cohort study will be conducted in women during pregnancy and lactation. From the first pregnancy visit until the child is six months old. Three prospectives (three annual series).

At least 60 healthy pregnant women and 60 women with a history of risk (20 for each risk) x 2 series (three years) will be tested, a total of 240-300 women to whom 5 analytical tests would have to be performed.

The researchers will take samples from the breastfeeding workshop of the study groups: Group 1 of healthy women and Group 2 of women with a history of risk (diabetes, overweight / obesity and hypertension)

DETAILED DESCRIPTION:
The project that is presented to the ethical committee, from the initial program called BECOME (Behavior of biomarkers (lipid profile and prolactin) during pregnancy and lactation through a biological multi-paradigm model), which already requested and obtained the Suitability dated April 28, 2015. Based on it, the development of the current project will be the historical memory of FPU Research Fellow (October 2016) The determination of the lipid profile in pregnancy is performed through blood tests in each of the quarters.

A prospective cohort study will be conducted in women during pregnancy and lactation. From the first pregnancy visit until the child is six months old. Three prospectives (three annual series).

At least 60 healthy pregnant women and 60 women with a history of risk (20 for each risk) x 2 series (three years) will be tested, a total of 240-300 women to whom 5 analytical tests would have to be performed.

The researchers will take samples from the breastfeeding workshop of the study groups: Group 1 of healthy women and Group 2 of women with a history of risk (diabetes, overweight / obesity and hypertension) Once all the data have been analyzed, a biological predictive model will be developed to establish its relationship with maternal alterations during pregnancy, as well as its relationship with lactogenesis in the last days of pregnancy. To this end, a computer program will be created where the personal, clinical and triglyceride levels of the pregnant woman will be obtained the results of the risk of altered triglycerides in the different months of gestation and the measures to be taken as a function of The same, as well as to identify the levels of triglycerides in the different maternal pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman with single pregnancy
* Pregnant woman with no assisted reproduction
* Pregnant woman from 12-14 weeks of gestation.

Exclusion Criteria:

* Pregnant woman with difficulty understanding the Spanish language
* Pregnant woman who have been diagnosed clinically of a chronic disease prior to pregnancy
* Pregnant woman who are under medical treatment (cancer, lung, kidney diseases , Hepatic, etc.).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Measurement of biomarker prolactin. | 10 months
  2- 6 days of delivery: Samples of: Colostrum. 7 to 21 days: Transition milk samples. From day 21: Sample of mature milk.
  For each of the above samples, it will be determined:
  * LIPIDIC PROFILE Short Chain Fatty Acids
  * Profile (quantification) of Total Fatty Acids. COMPLEMENTARY PARAMETERS: TG, Cholesterol, and Glucose, by R-Biopharm® Enzyme Test.
  Prolactin
Measurement of biomarker lipids | 10 months
  A test that measures the amount of lipids, or fat, in the blood. The lipids measured are: total cholesterol, HLD cholesterol, LDL cholesterol, and triglycerides.
  Laboratory diagnostic performance (hypertriglyceridemia)
  * Cholesterol, triglycerides, HDL cholesterol and non-HDL cholesterol
  * Glucose, creatine, ALT, GGT, uric acid, TSH
  * Sedimentation and semiquantitative proteinuria. Album / creatine ratio
  * Apolipoprotein B
  * Genotype of apolipoprotein E

SECONDARY OUTCOMES:
Anthropometric study. | 10 months
  Weight.- Size.- Seated size.- Triceps fold.- Biceps fold. -Subescapular fold.- Fold of ileocrestal.- Supraspinal fold.- Abdominal fold.- Axillary fold.-Folding pectoral.- Folding thigh frontal.- Fold leg Medial (calf) .- Perimeter of the relaxed arm.- Perimeter of the contracted arm.- Medial thigh perimeter.- Perimeter of the calf.- Diameter of the humerus.- Diameter of the wrist.- Diameter of the femur.- Diameter of the ankle
nutritional study. | 10 months
  For the study of the diet will be used 3 types of questionnaires:
  * Food register, in which the patient must record prior weighing or measurement, each and every one of the foods eaten during the day.
  * Reminder Questionnaire 24 hours. By means of which, the interviewer will ask the patient everything she has eaten the day before, and the quantities ingested, for which it will be used a photo album of weights and rations prepared by professors of the Department of Nutrition and Bromatology of the Faculty of Pharmacy
  * Frequency questionnaire of food consumption. By which the patient will indicate the times to the day, to the week, to the month or to the year that has consumed the food in the collected
Family history of illness. | 10 months
  Compiled from clinical history
demographic variables | 10 months
  Compiled from clinical history
Personal history of illness. | 10 months
  Compiled from clinical history

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granda, Granada, Spain